CLINICAL TRIAL: NCT07071857
Title: Coronary Artery Bypass Grafting With Concomitant Ascending Aortic Replacement: a Case-control Study
Brief Title: Coronary Artery Bypass Grafting With Ascending Aortic Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tomsk Cardiology Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CASE
Record Dates: First submitted 2025-07-04; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Coronary Artery Disease; Ascending Aortic Aneurysm
Keywords: CABG; ascending aortic aneurysm; aortic replacement; TTFM; MACCE
MeSH Terms: conditions — Coronary Artery Disease; Aneurysm, Ascending Aorta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CABG (Coronary artery bypass grafting) (Experimental): 35 patients who underwent isolated coronary artery bypass grafting.
  Interventions: Diagnostic Test: ECG CT angiography; Diagnostic Test: TTFM; Diagnostic Test: computed tomography of the aorta and/or grafts
- CABG+AAR (Coronary artery bypass grafting concomitant with ascending aortic replacement) (Experimental): 35 patients who underwent CABG concomitant with ascending aortic replacement.
  Interventions: Diagnostic Test: ECG CT angiography; Diagnostic Test: TTFM; Diagnostic Test: computed tomography of the aorta and/or grafts

INTERVENTIONS:
Diagnostic Test: ECG CT angiography — Preoperative: electrocardiography-gated computed tomographic angiography.
Diagnostic Test: TTFM — Intraoperative: TTFM after weaning from cardiopulmonary bypass and just before sternal closure.
Diagnostic Test: computed tomography of the aorta and/or grafts — computed tomography of the aorta and/or grafts within 2 weeks after surgery.

SUMMARY:
This retrospective study investigates early outcomes after CABG as well as graft patency rate in patients with concomitant AAR. 35 patients undergoing CABG with concomitant AAR (CABG+AAR group) were case-control matched to 35 patients who received isolated CABG (CABG group) in regard to transit-time flow measurement (TTFM) findings, early and late outcomes.

DETAILED DESCRIPTION:
1. Relevance of the study. Coronary artery bypass grafting is an effective treatment for patients with coronary artery disease (CAD). Nowadays, this operation is the most common surgical procedure performed on the heart, with >600,000 operations per year worldwide. Approximately 15-20% of patients with CAD require concomitant cardiac surgery with relatively high incidence of postoperative morbidity and mortality. It is considered that concomitant CAD in patients undergoing thoracic aortic surgery is an independent risk factor for perioperative mortality. Taking into account the recently published data, CABG added to other cardiac surgeries is associated with increased short- and long-term mortality. There are no available data on the relationship between the outcomes of the concomitant CABG and the patency of coronary grafts. The aim of this study was to assess the early outcomes after CABG as well as graft patency rate in patients with concomitant AAR.
2. Patients and methods. 35 patients who underwent CABG concomitant with ascending aortic replacement (CABG+AAR group) were compared with 35 patients who underwent isolated CABG (CABG group). Baseline characteristics which included preoperative characteristics, details on surgery (duration of cardiopulmonary bypass, cardioplegic arrest, antegrade cerebral perfusion), and early and late postoperative outcomes were compared between these groups.

Imaging All aortic measurements and postoperative graft patency were assessed by electrocardiography-gated computed tomographic angiography. Postoperative computed tomography of the aorta and/or grafts was performed within 2 weeks after surgery. Analysis was performed using 64-slice scanner Discovery NM-CT 570c (GE Healthcare, Milwaukee, WI, USA) with spatial resolution of the angiographic phase ranging from 0.6 to 1.25 mm. All measurements were taken always in the plane perpendicular to the manually corrected local aortic centre line. Ascending aortic diameter was measured at the level of the pulmonary artery bifurcation. The maximum aortic diameter (mm) was measured from the outer contours of the aortic wall.

The postoperative graft status was classified according to Fitzgibbon classification where Grade A is a patent graft, grade B is a stenosed graft (<50% of the grafted coronary artery) or a string sign and grade O is an occluded graft. All images were independently assessed by two experienced cardiologists.

Surgical technique CABG surgery was performed in the standard manner with a cardiopulmonary bypass and carioplegic arrest. Left internal mammary arterial (LIMA) grafts were used as in situ grafts to the LAD in all of the cases. All saphenous vein grafts (SVGs) were used in an aortocoronary bypass fashion. Proximal anastomoses were sewn to the aorta/graft with side-biting clamp on the beating heart.

The surgery was performed through a median sternotomy under mild-to-moderate hypothermia (28-30°C) and antegrade cerebral perfusion via the innominate artery with side graft. The distal aortic anastomosis was performed using an open anastomosis fashion and involved resection of the inferior portion of the aortic arch from the base of the innominate artery to the projection of the origin of the left subclavian artery (hemiarch repair). Near infrared spectroscopy (Invos 5100, Somanetics Corp., USA) was used for cerebral monitoring during the operation. When the target temperature was achieved, lower body circulatory arrest with antegrade cerebral perfusion was initiated. The distal aortic anastomosis was performed with a running 4/0 polypropylene suture with a Dacron graft. Proximal aortic anastomosis as well as coronary artery bypass grafting was performed during the rewarming period. The patient was weaned from cardiopulmonary bypass when the body temperature reached 36°C. The sequence of the surgical steps during the operation was the same for all patients.

Transit time flow measurement Graft flow tracing was recorded intraoperatively after weaning from cardiopulmonary bypass and just before sternal closure with a transit-time flowmeter (VQ1001, Medi-Stim AS, Oslo, Norway). The haemodynamic condition remained stable with a mean blood pressure between 70 and 90 mmHg during the flow measurement. The device displays a flow curve and calculates the mean graft flow (MGF) (ml/min), pulsatile index (PI) and diastolic filling percentage (DF%). The TTFM criteria for graft revision were MGF of <5 ml/min, PI of >5 or DF ratio of <50%.

Follow-up Follow-up was performed according to the institutional database supplemented by individual patient records. Data was obtained via medical records of clinical encounters or phone calls with patients and/or relatives. Postoperative computed tomographic scans and angiograms were performed upon discharge, at 12 months from the last procedure and annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years.
2. Signed informed consent.
3. Severe left main stem artery stenosis, or left main equivalent disease (70% or greater stenosis in diameter of the left anterior descending artery, proximal left circumflex artery and right coronary artery).
4. Ascending aorta greater than 5 cm.

Exclusion Criteria:

1. Dissections or urgent/emergent cases.
2. Redo aortic surgery.
3. Total aortic arch surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-01-20 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
major adverse cerebral and cardiac events (MACCE). | 12 months
  The difference in the incidence of MACCE between groups (p-value)

SECONDARY OUTCOMES:
Respiratory failure (%) | Perioperative
  The difference in the incidence of respiratory failure (p-value)
Acute kidney injury requiring renal replacement therapy (%) | Perioperative
  The difference in the incidence of renal replacement therapy during follow-up (p-value)
Re-exploration rate (%) | Perioperative
  The difference in the incidence of re-operation for bleeding during follow-up (p-value)

CONTACTS AND LOCATIONS:
Overall Officials: Boris N. Kozlov, MD, PhD, Principal Investigator — Cardiology Research Institute, Tomsk National Research Medical Center

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data (text, tables, figures, and appendices), underlying the results of the trial, will be shared with researchers to achieve the aims in the approved proposal
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Proposals may be submitted up to 36 months following publication of the results of the trial. After 36 months, the data will be available in the Center's data ware house but without investigator support other than deposited metadata
Access Criteria: Information regarding submitting proposals and accessing data may be requested from the principal investigator by e-mail.